CLINICAL TRIAL: NCT06397495
Title: Comparison of Flipped and Team-Based Learning Models in Cervical Region Manual Therapy Teaching: A Mixed Method Study
Brief Title: Comparison of Learning Models in Physical Therapy Education
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isparta University of Applied Sciences (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other); Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Ziya Yildiz, Expert Physiotherapist, Isparta University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SülDemirelUni_YildizZ_001
Record Dates: First submitted 2024-04-25; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Educational Problems; Surveys and Questionnaires
Keywords: Flipped Model; Physiotherapy Education; Cervical Manual Therapy; Psychomotor Skill
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flipped Groups (Experimental)
  Interventions: Other: Education
- Traditional Learning Groups (No Intervention)

INTERVENTIONS:
Other: Education — Cervical region manual therapy training will be given with flipped learning models.
  Arms: Flipped Groups

SUMMARY:
With the pandemic affecting the world, education systems have been subjected to mandatory changes without sufficient thought on teaching content, delivery and pedagogy. In this process, physiotherapy courses involving psychomotor skills such as manual therapy became difficult to teach and evaluate. Although the pandemic is over, it is suggested that technological approaches should be used in learning systems and incorporated into physiotherapy education. These technology-supported education models are called blended education models. The use of the flipped training model, a variant of blended training models, can improve practical skill performance. In this study, it was aimed to determine the effect of two different models on the quality of teaching and learning in cervical region manual therapy teaching. Suleyman Demirel University Physiotherapy and Rehabilitation senior students (n=100) will be randomly divided into two groups. The control group (n=49) will be given monologue education with in-class team-based traditional education model. The practical part of the course will be taught in the classroom and applied with patient-clinician role model technique. Homework will be assigned for students to read scientific articles and analyze case examples. The entire six-week teaching program will take place in the classroom. The experimental group (n=51) will be applied the flipped model. The theoretical and practical knowledge of the course will be provided at home with the EdPuzzle education platform. They will be encouraged to read articles and analyze cases at home. The classroom environment will be used to ask questions related to the theoretical part of the course and to practice the practical application as a patient/clinician role model. The seven-week teaching program is planned in the classroom and home environment. In the evaluation of the research, explanatory sequential design method from mixed research methods will be applied. Pre-test/post-test/knowledge retention test, instructional materials motivation questionnaire and skill level/performance evaluation form will be used to evaluate the quantitative data. A lesson observation form will be used to evaluate whether the trainer provided the same competence to both groups. Semi-structured case study will be used to evaluate the reverse-face model to the experimental group with qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* Not to have participated in a vocational course program on manual therapy of the cervical region,
* Sufficient internet access,
* Acceptance of distance education if included in the experimental group,
* Having and actively using a cell phone or computer with a smart operating system,
* Volunteering to participate in the study

Exclusion Criteria:

* The student wants to quit the study and does not fill in the data collection forms

Ages: 21 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2024-05-27 (Estimated)

PRIMARY OUTCOMES:
Academic motivation survey data | 1 year
  Academic motivation survey data will be the first data to be obtained between the groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Süleyman Demirel Univesity, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided